CLINICAL TRIAL: NCT05756296
Title: The Long-term Consequences of Neonatal Encephalopathy in the Hypothermia Era: Protocol for a Follow-up Cohort Study at 9 Years of Age
Brief Title: The Long-term Consequences of Neonatal Encephalopathy in the Hypothermia Era
Status: Not yet recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Marie Brossard-Racine, Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: MP-37-2023-9320
Record Dates: First submitted 2023-02-14; First posted 2023-03-06 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Neonatal Encephalopathy; Therapeutic Hypothermia; Brain Injuries; Child Development
Keywords: Cerebral Palsy; Brain; Neonate; Developmental Delay; MRI; Child Development
MeSH Terms: conditions — Brain Injuries; Cerebral Palsy; Learning Disabilities | interventions — Hypothermia, Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: Children aged 9 years old with NE-TH meeting study inclusion criteria.
  Interventions: Procedure: Therapeutic hypothermia
- Control group: A comparison group of sex and age matched children with no NE-TH meeting similar study inclusion criteria to intervention group. Specific exclusion criteria for matched control group include a previous history of neurodevelopmental delay or disorder, or a traumatic brain injury, and born at term (gestational age ≥37 weeks), or born without neonatal complication.

INTERVENTIONS:
Procedure: Therapeutic hypothermia — whole-body cooling to an esophageal temperature of 33.5°C initiated within the first 6 hours of life, continued for 72 hours, and then they were slowly rewarmed for moderate or severe NE
  Groups: Intervention group

SUMMARY:
The goal of this study is to characterize the ability and related brain profiles of children with Neonatal encephalopathy (NE) - Therapeutic hypothermia (TH) at 9 years old. The main questions it aims to answer are:

1. Compare executive function, attention, social cognition, behaviour, anxiety, self-esteem, and peer problems between children with NE-TH and matched peers without NE.
2. Compare brain volumes, cortical and subcortical morphology, white matter microstructure, and myelination between children with NE-TH and matched peers without NE.
3. Evaluate the associations of perinatal risk factors and structural brain integrity with neuropsychological deficits to inform about the potential aggravating and protective factors for neuropsychological functioning.

Participants will complete one study visit to perform standardized evaluations and a brain MRI. Parents of participants will be invited to complete a series of questionnaires during this study visit or at a moment of their choice virtually.

DETAILED DESCRIPTION:
Rationale:

Therapeutic hypothermia (TH) became the standard of care treatment for neonates with moderate and severe neonatal encephalopathy (NE) in most industrialized countries about 10 years ago. Although TH is effective in reducing mortality and the incidence of severe developmental disabilities, various morbidities are still frequent in survivors. Moreover, because the focus of previous follow-up studies has been restricted to mortality rates and the most severe forms of morbidities, it is wrong to conclude that TH minimizes all developmental deficits. In fact, recent literature reports frequent cognitive and behavioural difficulties at school entry in children with NE-TH without severe disabilities. Although these difficulties can be less impressive than cerebral palsy and intellectual disability, their negative impacts on a child's self-determination and family well-being are not less important and their nature and extend need to be comprehensively assessed.

Aims and Hypotheses:

1. To compare higher-order cognitive, socialization, and psycho-emotional abilities using comprehensive standardized assessments of outcomes between 9-year-old children with NE-TH and age- and sex-matched peers without NE.

   Hypothesis 1: Children with NE-TH will display lower IQ, executive functioning, attention, social cognition, and self-esteem, but more anxiety and behavioural and peer problems than age- and sex-matched peers without NE-TH.
2. To compare structural brain integrity using quantitative MRI between 9-year-old children with NE-TH and age- and sex-matched peers without NE.

   Hypothesis 2: Children with NE-TH will present with smaller total and regional (basal ganglia, hippocampus, cerebellum) brain volumes, altered cortical and subcortical morphometry, and widespread white matter microstructural and myelination alterations when compared to age- and sex-matched peers without NE-TH.
3. To evaluate the relationships between cognitive, psycho-emotional and motor skills at 9 years and (1) individual and perinatal risk factors and (2) structural brain integrity at 9 years.

Hypothesis 3: A combination of individual (e.g., socio-economic), perinatal factors (e.g., neonatal brain injury) and markers of aberrant brain integrity (e.g., volume, microstructure) will be associated with domain-specific deficits at 9 years in children with NE-TH.

Population:

Children born between 2014 and 2018, who received whole-body cooling to an esophageal temperature of 33.5°C initiated within the first 6 hours of life, continued for 72 hours, and then they were slowly rewarmed for moderate or severe NE at one of the two centers will be approached. Eligibility for TH at our institutions followed those established in previous TH trials. Participants with a history of (1) congenital infections, (2) genetic or metabolic disorders, or (3) major brain malformations (e.g., lissencephaly), as well as (4) any contraindication for MRI (e.g., metal implant, claustrophobia), are ineligible.

For each of two same-sex and same-age NE-TH participants, a matched control for age (+/- 6 months of mean age) and sex will be recruited. Participants born at term (gestational age ≥37 weeks), without neonatal complication, will be considered as ineligible controls. Inclusion criteria for the controls include the same were similar to the NE-TH group, and a previous history of neurodevelopmental delay or disorder, or a traumatic brain injury were the specific exclusion cirteria for the comparison group.

Assessment procedure:

For this study, enrollees will complete one study visit to perform standardized evaluations and a brain MRI. Children will have the opportunity to familiarize themselves with the MRI environment on a mock scanner before the MRI and to watch a movie or listen to the music of their choice during the acquisition. Parents will be invited to complete a series of questionnaires during their child's testing or at a moment of their choice via a provided secure link. The visit will start with the outcome evaluations that are the most cognitively demanding and breaks will be provided as necessary. Outcome evaluations will be conducted by trained research staff or trainees blinded to the details of the child's neonatal and developmental history, and group allocation (i.e., NE-TH vs. control) to the extent possible. The choice of outcome measures has been made based on their clinical significance, psychometric properties, and availability in both French and English, considering the bilingual context of Quebec, Canada.

ELIGIBILITY:
Inclusion Criteria:

* born between 2014 and 2018
* received whole-body cooling to an esophageal temperature of 33.5°C initiated within the first 6 hours of life, continued for 72 hours, and then they were slowly rewarmed received TH for moderate or severe NE

Exclusion Criteria:

Participants with a history of

* congenital infections
* genetic or metabolic disorders
* major brain malformations (e.g., lissencephaly) and
* any contraindication for MRI (e.g., metal implant, claustrophobia)

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Existing clinical cohort of children born between 2014 and 2018, who received TH for NE treated at the two largest neonatal intensive care units and neonatal follow-up programs in Quebec (Canada), the Montreal Children's Hospital (MCH) of the McGill University Health Centre and the Centre Hospitalier Universitaire Ste-Justine (CHUSJ).
Sampling Method: Non-Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Higher order cognitive abilities | DAY 1
  Estimated IQ (Wechsler Abbreviated Scale of Intelligence 2nd ed. [WASI-2]), inhibition (Stroop test), planning (Tower - Delis-Kaplan Executive Function System [D-KEFS] and Rey-Osterrieth Complex Figure), impulsivity (Conner Continuous Performance Test - 3rd Ed [CPT-3]), working memory (Digit span), and word retrieval (verbal fluency - D-KEFS). Specific attentional skills; immediate (Digit Span) and sustained attention (CPT-3). Visual memory (Rey-Osterrieth Complex Figure). To characterize the ability to understand that others have thoughts, ideas, and feelings, and how emotion relates to social context, as well as the ability to recognize affect (Theory of Mind and Affect Recognition subtests).
Psycho-emotional abilities | DAY 1
  Self-esteem (Self-Concept Inventory from the Beck Youth Inventories-II), children's anxiety and emotional regulation (Spence Children's Anxiety Scale, the Multidimensional Anxiety Scale for Children, and the Difficulties in Emotion Regulation Scales). Predominance of profiles (e.g., predominantly affective, cognitive, or generalized) will be examined following an in-depth interpretation of the cognitive and psycho-emotional outcomes.
Motor skills | DAY 1
  Motor skills will be evaluated using the Movement Assessment Battery for Children-2nd Ed.in children without CP. In children with CP, motor skills will be evaluated with the Gross Motor Function Measure and subsequently be classified using the Gross Motor Function Classification System and the Manual Ability Classification System.Visual-motor integration will be assessed with the Berry-Buktenica Developmental Test of Visual-Motor Integration.
Functional profile | DAY 1
  Adaptive Behaviour Assessment Systems 3rd Ed.
Brain profile | DAY 1
  Quantitative MRI measuring structural brain integrity

OTHER OUTCOMES:
Sex | DAY 1
  determined by the physical appearance of genitalia recorded at birth
Gender | DAY 1
  self-reported by the child
Socio-economic status | DAY 1
  Maternal Education, employment, income and ethnicity
Medical history of child | DAY 1
  prenatal, perinatal, and postnatal factors extracted from existing clinical and research databases

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Centre Hospitalier Universitaire Ste-Justine (CHUSJ)., Montreal, Quebec
  - the Montreal Children's Hospital (MCH) of the McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Background] Shankaran S, Laptook AR, Ehrenkranz RA, Tyson JE, McDonald SA, Donovan EF, Fanaroff AA, Poole WK, Wright LL, Higgins RD, Finer NN, Carlo WA, Duara S, Oh W, Cotten CM, Stevenson DK, Stoll BJ, Lemons JA, Guillet R, Jobe AH; National Institute of Child Health and Human Development Neonatal Research Network. Whole-body hypothermia for neonates with hypoxic-ischemic encephalopathy. N Engl J Med. 2005 Oct 13;353(15):1574-84. doi: 10.1056/NEJMcps050929. PMID 16221780
- [Background] Levine DS. Neuroexecutive Function. In: Encyclopedia of Human Behavior.2012:701-706
- [Background] Scarpina F, Tagini S. The Stroop Color and Word Test. Front Psychol. 2017 Apr 12;8:557. doi: 10.3389/fpsyg.2017.00557. eCollection 2017. PMID 28446889
- [Background] Deli DC, Kaplan E, Kramer JH. Delis-Kaplan Executive Function System. Pearson Publication Inc; 2001
- [Background] Rey A. L'examen psychologique dans les cas d'encéphalopathie traumatique. (Les problems.). [The psychological examination in cases of traumatic encepholopathy. Problems.]. Archives de Psychologie. 1941;28:215-285
- [Background] Conners CK. Conner Continuous Performance Test - 3rd Ed Pearson Publication Inc.; 2014.
- [Background] Hunt C, Borgida E, Lavine H. Social Cognition. In: Encyclopedia of Human Behavior.2012:456-462
- [Background] Korjman M, Kirk U, Kemp S. NEPSY Second Edition (NEPSY-II): A developmental NEuroPSYchological Assessment. Pearson Publication Inc; 2007
- [Background] Roid GH, Miller LJ. Leither Internaltional Performance Scale - Revised. Wod Dale, IL: Stoelting; 1997
- [Background] Thompson EJ, Beauchamp MH, Darling SJ, Hearps SJC, Brown A, Charalambous G, Crossley L, Darby D, Dooley JJ, Greenham M, Jaimangal M, McDonald S, Muscara F, Turkstra L, Anderson VA. Protocol for a prospective, school-based standardisation study of a digital social skills assessment tool for children: The Paediatric Evaluation of Emotions, Relationships, and Socialisation (PEERS) study. BMJ Open. 2018 Feb 8;8(2):e016633. doi: 10.1136/bmjopen-2017-016633. PMID 29439065
- [Background] Beck J, S., Beck A, T., Jolly J, B. . Beck Youth Inventories - Second Edition. San Antonio, TX: Peason; 2005
- [Background] Spence SH. Spence Children's Anxiety Scale. Washington, DC: American Psychology Association; 1997
- [Background] March JS, Parker JD, Sullivan K, Stallings P, Conners CK. The Multidimensional Anxiety Scale for Children (MASC): factor structure, reliability, and validity. J Am Acad Child Adolesc Psychiatry. 1997 Apr;36(4):554-65. doi: 10.1097/00004583-199704000-00019. PMID 9100431
- [Background] Gratz KL, Roemer L. Multidimensional Assessment of Emotion Regulation and Dysregulation: Development, Factor Structure, and Initial Validation of the Difficulties in Emotion Regulation Scale. Journal of Pyschopathology and Behavioral Assessment. 2004;26(1):41-54
- [Background] Russel DJ, Rosenbaum P, Wright M, Avery LM. Gross Motor Function Measure (GMFM-66 & GMFM-88) User's Manual, 2nd Edition. 2nd ed: Mac Keith Press; 2013
- [Background] Harrison P, Oakland T. Adaptive Behavior Assessment Systems 3rd Ed. Pearson Publication Inc; 2015.
- [Derived] Brossard-Racine M, Rampakakis E, Tardif CL, Gilbert G, White A, Luu TM, Gallagher A, Pinchefsky E, Montreuil T, Simard MN, Wintermark P. Long-term consequences of neonatal encephalopathy in the hypothermia era: protocol for a follow-up cohort study at 9 years of age. BMJ Open. 2023 Apr 13;13(4):e073063. doi: 10.1136/bmjopen-2023-073063. PMID 37055215